CLINICAL TRIAL: NCT06755801
Title: Microvascular Obstruction Treatment and Outcomes Randomized Study.
Brief Title: Nebivolol ANOCA Treatment Randomized Trial
Acronym: MOTORS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Fernando Alfonso, Head of Cardiology Department. H. U. de la Princesa., Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sec1589634
Record Dates: First submitted 2024-12-06; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: ANOCA - Angina With Non-obstructive Coronary Arteries; Coronary Microvascular Dysfunction (CMD)
Keywords: Coronary Microvascular Disease; Betablockers; Angina
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment group (Experimental): Nevibolol tratment
  Interventions: Drug: Nevibolol
- Control group (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nevibolol — Beta-blockers are the first-line treatment for patients with stable angina secondary to classic epicardial atherosclerotic disease, where their clinical benefits are well-established (4). However, their efficacy has not yet been demonstrated in ANOCA patients with MVD, where beta-blockers are frequently used due to their physiological plausibility. Beta-blockers act by competitively inhibiting catecholamine receptors. The therapeutic benefits of beta-blockade in patients with stable angina are mediated by a reduction in myocardial oxygen demand. Myocardial oxygen demand depends on heart rate, contractility, and left ventricular wall tension, all of which are reduced with beta-adrenergic blockade. The reduction in wall tension is partly mediated by the antihypertensive action of these drugs. The decrease in heart rate occurs both at rest and during sympathetic activation such as exercise or stress. The negative inotropic effect of these drugs also contributes to reducing myocardial oxyg
  Arms: Active treatment group
Drug: Placebo — Placebo
  Arms: Control group

SUMMARY:
To determine the effectiveness of the beta-blocker nebivolol in controlling symptoms and improving the quality of life in patients with angina and coronary microvascular dysfunction.

DETAILED DESCRIPTION:
Objective To determine the effectiveness of the beta-blocker nebivolol in controlling symptoms and improving the quality of life in patients with angina and coronary microvascular dysfunction.

Hypothesis Treatment with titrated nebivolol will result superior to placebo in symptoms control in patients presenting with coronary microvascular disease (CMD).

Study design Prospective, multicenter, controlled, double-blinded, randomized clinical trial.

Inclusion criteria • Patients over 18 years old with symptoms or evidence of myocardial ischemia and coronary arteries without lesions or with epicardial lesions (<50% by visual estimation or FFR >0.80 / RFR >0.90), and

• CFR ≤ 2.0 and/or IMR≥25 Exclusion criteria Life expectancy <1 year, inability to provide informed consent, severe valve disease, left ventricular ejection fraction <30%, clinical contraindication for betablockers treatment.

Treatment arms Randomization will be performed after invasive diagnostic of CMD:

Study group: Nebivolol • Patients will start with a dose of 5 mg every 24 hours. Biweekly dose adjustments will be performed during the first two months, increasing the dose (if tolerated with respect to heart rate, blood pressure, and symptoms) up to a maximum of 20 mg/24 hours.

Control group: Placebo

• Patients will be treated with one tablet every 24 hours. Primary endpoint: The effectiveness of nebivolol treatment in improving angina symptoms was measured using the SAQ questionnaire after 6 months of treatment.

Secondary endpoints • Quality of life at 6 months.

* Functional capacity at 6 months.
* Major cardiac events at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.

  * Presence of stable angina symptoms, defined as compatible symptoms occurring at least once weekly in the last three months.
  * Absence of functionally significant epicardial coronary artery disease (FFR > 0.80).
  * Microvascular functional study showing CFR< 2,0 and/or IMR ≥ 25.

Exclusion Criteria:

* Allergy or contraindication to the use of beta-blockers.
* Indication for beta-blocker treatment due to another pathology.
* Ventricular dysfunction (LVEF < 45%).
* Percutaneous coronary revascularization in the last 6 months.
* History of surgical revascularization.
* First-degree atrioventricular block or bifascicular block.
* Presence of hemodynamically significant valvulopathy.
* Presence of cardiomyopathy or congenital cardiac anomaly.
* Severe renal insufficiency (eGFR < 30 ml/min).
* Liver failure (history of cirrhosis or transaminase elevation > 3 times the upper limit of normal).
* Pregnant or lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
SAQ questionnaire | 6 months
  The pre-specified primary outcome criterion is the improvement in angina severity assessed by the Seattle Angina Questionnaire (SAQ SS - Summary Score) at 6 months from the start of treatment compared to baseline. It will be evaluated by the mean difference in change within the same patient in SAQ between the two groups at 6 months of treatment.
  The SAQ is a validated self-administered scale that allows assessment of angina severity, frequency, quality of life, and functional limitation. It is the most commonly used and validated patient-reported outcome measure for angina. The SAQ provides a scale for evaluating the severity of angina that has been shown to be valid, reproducible, and sensitive to changes.

SECONDARY OUTCOMES:
Quality of Life Status using the EuroQOL questionnaire (EQ5D-5L) | 6 months
  Patient's quality of life in both treatment groups will be assessed using the EuroQOL questionnaire (EQ5D-5L). The EQ5D-5L is the most widely used instrument for assessing health-related quality of life.
the Brief Illness Perception Questionnaire (B-IPQ) | 6 months
  Changes in disease perception will also be recorded using the Brief Illness Perception Questionnaire (B-IPQ)
anxiety and depression using PHQ-4 | 6 months
  Quality of Life Status
The treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM-9) | 6 months
  Quality of Life Status
Functional Capacity | 6 months
  Functional capacity in both groups will be objectively assessed by performing a baseline and 6-month exercise treadmill test (ergometry) according to the Bruce protocol. The evaluated parameter will be the total duration of maximum exercise (seconds).
Major Cardiac Events | 6 months
  The presence of major cardiac events will be adjudicated by an Independent Events Committee. Major cardiac events are defined as death from any cause, acute myocardial infarction, and hospitalization due to unstable angina, stroke, or heart failure requiring hospitalization.

IPD SHARING:
Plan to Share IPD: Undecided